CLINICAL TRIAL: NCT01429012
Title: Treatment of Atrophic Nonunion Fractures by Autologous Mesenchymal Stem Cell Percutaneous Grafting. A Randomized, Double-blind, Controlled Study
Brief Title: Treatment of Atrophic Nonunion Fractures by Autologous Mesenchymal Stem Cell Percutaneous Grafting
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Yves Beguin, MD, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJT1101
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Nonunion Fracture
Keywords: bone; nonunion fracture; atrophic nonunion fracture; callus; mesenchymal stem cells; cell therapy; autologous; indium; Pet-scan
MeSH Terms: conditions — Fractures, Ununited; Callosities | interventions — Culture Media

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesenchymal Stem Cells (Experimental): 2 ml with 40 X 10E6 Mesenchymal Stem Cells (MSC) will be injected in the nonunion space of the bone fracture.
  MSC will be injected even if the number of available cells is lower than 40 X 10E6.
  The injection of MSC in the nonunion space will be performed percutaneously using a 3-mm trephine needle under fluoroscopic control and loco-regional or general anesthesia, as deemed appropriate by the anesthetist.
  Interventions: Biological: Mesenchymal Stem Cells
- Culture medium without MSC. (Placebo Comparator): Culture medium used to resuspend the Mesenchymal Stem Cells.
  Interventions: Other: Culture medium without MSC.

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — Mesenchymal Stem Cells. Dose= 40 X 10E6 in 2 ml. Frequency = one injection. If no evidence of a callus after 6 months a second injection can be proposed.
  Other Names: MSC
  Arms: Mesenchymal Stem Cells
Other: Culture medium without MSC. — 2 ml of culture medium.
  Arms: Culture medium without MSC.

SUMMARY:
Bone fractures heal most of the time particularly well and without complications. The solidification takes rarely more than two to three months. The wound healing depends greatly on a good blood supply and needs several steps. These processes culminate in a new mass of heterogeneous tissue which is known as the fracture callus. Unfortunately, 2%-5% bone fractures cannot achieve a proper solidification and between the ununited fragments a scar tissue appears. This incorrect healing induces pain and even infections. When this situation persists more than 6 months, it is referred to as nonunion fracture, which will require some form of intervention to stimulate the natural healing process of the body. First of all, good surgical techniques with stable immobilization should be applied and local infection should be excluded. Then stimulation of the callus is required. Cell therapy with bone marrow cells has emerged as a promising new approach for bone regeneration. Animal studies as well as preliminary human studies have shown that Mesenchymal Stem Cells, a particular kind of stem cells isolated from the bone marrow, could induce callus formation when injected in the nonunion site of a broken bone.

In this study the investigators aim at determining whether Mesenchymal Stem Cells (MSC) isolated from the patient's bone marrow and injected in the nonunion site could be a safe and effective treatment for nonunion fractures. Patients will be randomized in two groups; one injected with Mesenchymal Stem Cell and the other injected with placebo. The investigators seek also to know how long it takes to develop the callus formation and whether there is a partial or a complete callus formation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; female patients must use a reliable contraception method
* Age ≥ 18 years
* Fracture having no radiological callus after 6 months and absence of any hypertrophic bone reaction.
* No sepsis
* Good skin covering
* Be able and willing to participate in the study
* Written informed consent

Exclusion Criteria:

* Evidence of malignancy (except non-melanoma skin cancer) in the past five years
* Pregnancy or breastfeeding
* Patient positive by serology or PCR for HIV, hepatitis B or C infection
* Insufficient reduction of the fracture with displaced fragments
* Evidence of local sepsis by clinical signs, biological parameters (CRP) and/or positive isotopic scan using Indium-labelled leucocytes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11 (Estimated); Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Safety of Mesenchymal Stem Cells injection in nonunion fractures. | 12 months
  Follow-up for revealing any significant immediate or late adverse effects.
Proportion of patients receiving Mesenchymal Stem Cells that develop a partial or complete callus at 6 and 12 months, compared to patients receiving placebo. | 6 and 12 months
  Radiological evaluation of the callus by standard X-rays and computed tomography (CT).

SECONDARY OUTCOMES:
Proportion of patients receiving Mensechymal Stem Cells that develop a partial or complete callus at 2, 3, 4, 8 and 10 months, compared to patients receiving placebo | 2, 3, 4, 8 and 10 months
  Radiological evaluation of the callus by standard X-rays and computed tomography (CT).
Timing of development of a partial or complete callus in the 2 groups. | 12 months for one injection or 18 months when a second injection is needed
  Time necessary for a partial or a complete callus formation. Radiological evaluation of the callus by standard X-rays and computed tomography (CT).
Patient evaluation of pain and global satisfaction. | 12 months
  This evaluation will be measured through a 100-mm Visual Analogue Scale at 2, 3, 4, 6, 8, 10 and 12 months in the 2 groups.
Proportion of patients achieving different degrees of functional success. | 2, 3, 4, 6, 8, 10 and 12 months
  The functional assessment will be evaluated in Mesenchymal Stem Cells treated and untreated patients by an orthopaedic surgeon and will include a 4-points scale:
  * 0 = only passive motion allowed
  * 1 = only active mobilization without any opposition allowed
  * 2 = active mobilization with some opposition and partial weight-bearing allowed
  * 3 = weight-bearing and full active mobilization allowed
Incidence of adverse events and severe adverse events in the 2 groups. | 12 months for one injection and 18 months when a second injection is performed
  Adverse events and serious adverse events will be continuously monitored .
Evaluation of early homing of Mesenchymal Stem Cells. | 24 hours
  Indium radiolabeled Mesenchymal Stem Cells (MSC) will be visualized with a Siemens e-CAM dual head gamma camera: 10% of the total amount of MSC will be incubated with 200 µCi In-111-oxine. The radiolabelled cells will be mixed with the unlabelled ones. Twenty-four hours after injecting the cells into the target bone lesion, static images centered over the injection site and whole-body images will be acquired during 20 minutes. This will be performed with a Siemens e-CAM dual head gamma camera.
Value of [18F]-NaF PET scans for early prediction of the onset of the bone healing process. | 3 months
  PET Fluor kinetics could identify early and perhaps quantify the increase of bone forming in the treated area. Four [18F]-NaF PET scan studies will be performed: at baseline, as well as around days 7-9 (1 week), 27-33 (one month) and 83-97 (three months).

CONTACTS AND LOCATIONS:
Overall Officials: Jean Philippe Hauzeur, MD, PhD, Principal Investigator — University of Liege; Yves Beguin, Prof, MD, PhD, Study Chair — University of Liege
Locations (1):
- Liège University Hospital, Liège, Belgium